CLINICAL TRIAL: NCT00612183
Title: Phase II Clinical Study on SyB L-0501 in Patients With Indolent B-cell Non-Hodgkin's Lymphoma or Mantle Cell Lymphoma (Multicenter, Open-label Study)
Brief Title: Clinical Study on SyB L-0501 in Patients With Indolent B-cell Non-Hodgkin's Lymphoma or Mantle Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SymBio Pharmaceuticals (Industry)
Responsible Party: Katsuhisa Goto, SymBio Pharmaceuticals Limited
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007002
Record Dates: First submitted 2008-01-28; First posted 2008-02-11 (Estimated); Last update posted 2010-07-22 (Estimated); Status verified 2010-05

CONDITIONS: Non-Hodgkin's Lymphoma; Mantle Cell Lymphoma
Keywords: non-Hodgkin's lymphoma; mantle cell lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Mantle-Cell | interventions — Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: bendamustine hydrochloride — bendamustine hydrochloride is administered by 60-min drip infusion at 120 mg/m2/day for 2 consecutive days, and the course is then observed for 19 days. This is one cycle and administration is repeated for 3 - 6 cycles. From the second cycle, the dose is reduced or administration is discontinued as required based on adverse events observed in the previous cycle or observation of the course.

SUMMARY:
The purpose of this study is to assess the antitumor effects and safety of bendamustine hydrochloride (SyB L-0501) in patients with indolent B-cell non-Hodgkin's lymphoma or mantle cell lymphoma.

DETAILED DESCRIPTION:
Indolent B-cell Non-hodgkin's lymphoma is treated mainly with radiation and chemotherapy using a combination of chemotherapies, such as purine-analogues and CHOP (cyclophosphamide, doxorubicin, vincristine and prednisolone). After the approval of an antibody therapy agent Rituximab®, it alone or combination with CHOP has been introduced. Bendamustine hydrochloride has a unique structure compared with the marketed agents, and has an innovative mechanism of action. Thus, it is expected that Bendamustine hydrochloride will provide new alternatives for patients with refractory/recurrent indolent B-cell Non-hodgkin's lymphoma.

ELIGIBILITY:
Inclusion Criteria:

Non-Hodgkin's lymphoma patients with prior therapy who satisfy the conditions listed below. No restrictions regarding gender.

* Patients with histologically or cytologically confirmed indolent B cell Non-Hodgkin's lymphoma or mantle cell lymphoma.
* Patients who had not received treatment for at least 4 weeks (for at least 12 weeks in the case of antibody therapy) after completion of prior therapy and who are judged to carry no effect from the prior therapy.
* Patients aged from 20 to less than 75 years.
* Performance Status (P.S.): 0 or 1.
* Patients with adequately maintained organ functions (e.g., bone marrow, heart, lung, liver, and kidney functions).
* Patients from whom written consent to participate in this study has been obtained.

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded.

* Patients with apparent infections.
* Patients with serious complications (hepatic failure or renal failure).
* Patients with complication or history of serious heart failure (e.g. cardiac infarction, ischemic heart disease).
* Patients with serious digestive symptoms (nausea/ vomiting/ diarrhea).
* Patients who are known to be positive for HBV, HCV or HIC.
* Patients receiving other investigational drugs within 3 months before registration in the study.
* Patients with allogenic bone-marrow transplant.
* Women who are pregnant, of childbearing potential, or lactating.
* Patients who do not agree to contraception.
* Otherwise, patients who are judged by the investigator as being unsuitable for inclusion in the study.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2007-12; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Overall response rate based on [Report of an International Workshop to Standardize Response Criteria for Non-Hodgkin's Lymphomas] | [Treatment period]

SECONDARY OUTCOMES:
CR rate of overall results based on [Report of an International Workshop to Standardize Response Criteria for Non-Hodgkin's Lymphomas] | [Treatment Period]

CONTACTS AND LOCATIONS:
Overall Officials: Kensei Tobinai, MD, PhD, Study Chair — National Cancer Center Hospital
Locations (17):
- Japan (17):
  - Nagoya, Aichi-ken
  - Kashiwa, Chiba
  - Fukuoka, Fukuoka
  - Sapporo, Hokkaido
  - Kagoshima, Kagoshima-ken
  - Isehara, Kanagawa
  - Kumamoto, Kumamoto
  - Kyoto, Kyoto
  - Sendai, Miyagi
  - Nagoya, Nagoya
  - Moriguchi, Osaka
  - Hamamatsu, Shizuoka
  - Utsunomiya, Tochigi
  - Chūō, Tokyo
  - Koto, Tokyo
  - Shibuya City, Tokyo
  - Shinagawa, Tokyo

REFERENCES:
- [Derived] Ohmachi K, Ando K, Ogura M, Uchida T, Itoh K, Kubota N, Ishizawa K, Yamamoto J, Watanabe T, Uike N, Choi I, Terui Y, Usuki K, Nagai H, Uoshima N, Tobinai K; Japanese Bendamustine Lymphoma Study Group. Multicenter phase II study of bendamustine for relapsed or refractory indolent B-cell non-Hodgkin lymphoma and mantle cell lymphoma. Cancer Sci. 2010 Sep;101(9):2059-64. doi: 10.1111/j.1349-7006.2010.01635.x. PMID 20626754